CLINICAL TRIAL: NCT06064071
Title: Clinical Study Evaluating Nordlys™ SWT IPL for Dry Eye Disease (DED) Due to MGD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DED23001
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Disease
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: Nordlys SWT IPL (Experimental): Subjects will receive up to four study Nordlys SWT IPL treatments and MGX
  Interventions: Device: Nordlys SWT IPL; Procedure: Meibomian Gland Expression (MGX)
- Control Group: Sham Treatment (Sham Comparator): Subjects will receive up to four sham study Nordlys SWT IPL treatments (device turned off) and MGX
  Interventions: Procedure: Meibomian Gland Expression (MGX); Device: Sham Nordlys SWT IPL

INTERVENTIONS:
Device: Nordlys SWT IPL — Nordlys™ System with Selective Waveband Technology (SWT)® IPL Applicators
  Arms: Experimental: Nordlys SWT IPL
Procedure: Meibomian Gland Expression (MGX) — Meibomian glands are squeezed (by applying force on the inner and outer surfaces of the eyelid with a specially designed forceps, Q-tips, or fingers) in order to unclog obstructed glands and evacuate their content (the meibum), which in MGD is often viscous and thus causing obstruction
Device: Sham Nordlys SWT IPL — Sham treatment with Nordlys™ System with Selective Waveband Technology (SWT)® IPL Applicators device turned off
  Arms: Control Group: Sham Treatment

SUMMARY:
Clinical Study Evaluating Nordlys™ System with Selective Waveband Technology (SWT)® Intense Pulsed Light (IPL) Applicators for Dry Eye Disease (DED) due to Meibomian Gland Dysfunction (MGD).

DETAILED DESCRIPTION:
Subjects will be randomized 1:1 to an experimental study group and a sham comparator (control) group.

Subjects in the experimental group will receive four (4) IPL treatments and meibomian gland expression (MGX) at 2-week intervals. IPL pulses will be administered on the skin of the malar region and below the lower eyelids. Following IPL therapy, subjects will undergo MGX of both eyelids in both eyes. Subjects in the control group will receive the same treatment (IPL followed by MGX), except that the IPL administration will be performed with the device off (sham treatment). Follow-up visits will occur at 1 month and 3 months after the final treatment session. At the follow-up, the changes in the outcome measures will be evaluated and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects between 18 to 75 years of age with Fitzpatrick Skin Type I - VI.
* Able and willing to comply with the treatment/follow-up schedule and requirements comply with all study (protocol) requirements.
* Willingness to provide signed, informed consent to participate in the study
* Willing to have photographs and images taken of the treated areas to be used in evaluations, publications, presentations, and marketing materials
* Has Tear Breakup Time (TBUT) ≤ 7 seconds at screening/baseline
* Has Meibomian gland secretion score (MGS) ≤ 12 at screening/ baseline
* Has at least 5 non-atrophied meibomian glands and at least 50% of working meibomian glands in the lower eyelid at screening/ baseline
* Symptoms self-assessed using the OSDI questionnaire ≥ 23 at screening/ baseline

Exclusion Criteria:

* Contact lens wear within the month prior to screening
* Unwilling to discontinue use of contact lenses for the duration of the study
* Ocular surgery or eyelid surgery, within 6 months prior to screening
* Neuro-paralysis in the planned treatment area, within 6 months prior to screening
* Other uncontrolled eye disorders affecting the ocular surface, for example active allergies
* Current use of punctal plugs
* Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
* Uncontrolled infections or uncontrolled immunosuppressive diseases
* Subjects with ocular infections, within 6 months prior to screening
* Prior history of cold sores or rashes in the perioral area or in the planned treatment area that could be stimulated by light at a wavelength of 560 nm to 1200 nm, including: Herpes simplex 1 & 2, Systemic Lupus erythematosus, and porphyria unless treated following a prophylactic regimen per principal investigator discretion.
* Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
* Over exposure to sun, within 4 weeks prior to screening
* Use of prescription eye drops for dry eye, within 7 days prior to screening, excluding artificial tears and glaucoma drops
* Radiation therapy to the head or neck, within 12 months prior to screening
* Planned radiation therapy, within 8 weeks after the last treatment session
* Treatment with chemotherapeutic agent, within 8 weeks prior to screening
* Planned chemotherapy, within 8 weeks after the last treatment session
* New topical treatments within the area to be treated, or oral therapies, within 3 months prior to screening- except over-the-counter acetaminophen-based analgesics for pain management, new oral omega 3 fatty acid supplements and topical artificial tears
* Change in dosage of any systemic medication, within 3 months prior to screening
* Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up over the study period
* Legally blind in either eye
* History of migraines, seizures or epilepsy
* Facial IPL treatment within 12 months prior to screening
* Any thermal treatment of the eyelids, including Lipiflow, within 6 months prior to screening
* Expression of the meibomian glands, within 6 months prior to screening
* In either eye, moderate to severe inflammation of the conjunctiva, including: allergic, vernal or giant papillary conjunctivitis or severe inflammation of the eyelid, including: blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis
* Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy)
* Eyelid abnormalities that affect lid function in either eye, including: entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, and severe ptosis
* Any systemic condition that may cause dry eye disease, including: Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, and Sjögren's syndrome
* Unwilling or unable to abstain from the use of medications known to cause dryness (e.g., isotretinoin, antihistamines) throughout the study duration. Subjects must discontinue these medications for at least 1 month prior to the baseline visit.
* Any condition revealed whereby the investigator deems the subject inappropriate for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of Tear Breakup Time (TBUT) from baseline to 4-week follow-up | Baseline, 4-Week Follow Up (Week 10)
  The difference in the change of TBUT from Baseline to Follow-Up, between eyes in the study group and eyes in the control group. TBUT is measured in seconds. Improvement is defined as a positive change of TBUT from Baseline to Follow Up. Measurement of TBUT will be implemented using fluorescein ophthalmic strips. Three successive readings will be taken and averaged to a single value.

SECONDARY OUTCOMES:
Difference in change of self-assessed symptoms with the Ocular Surface Disease Index (OSDI) questionnaire, from baseline to follow-up. | Baseline, 1 Month Follow Up at Week 10, and 3 Month Follow Up at Week 18
  The difference in the change of OSDI from baseline to FU, between subjects in the study group and subjects in the control group. The minimal number is 0 and the maximal number is 100. Higher scores mean worse outcome. A score of 0-12 is considered normal. A score of 13-22 is consistent with mild dry eye. A score of 23 to 32 is consistent with moderate dry eye. A score from 33 to 100 is consistent with severe dry eye. The improvement of OSDI is defined as a negative change of OSDI from BL to FU.
The difference in change of self-assessed symptoms of eye dryness via Eye Dryness Score (EDS) via visual analog scale (VAS), from baseline to follow-up | Baseline, 1 Month Follow Up at Week 10, and 3 Month Follow Up at Week 18
  A qualitative test to visualize the production of sweat to the affected body area and assist in determining the area requiring treatment. Values will be collected separately for each eye. Correlation between eyes was removed by statistical methods. Scores were 0 (minimum) to 100 (maximum). Higher scores = worse outcome. The improvement of EDS is defined as a negative change of EDS from baseline to follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Center for Excellence in Eye Care, Miami, Florida
  - Candela Institute of Excellence, Marlborough, Massachusetts
- Av. Del Libertador 662, Piso 17, Dept. 42, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No